CLINICAL TRIAL: NCT04072900
Title: A Phase I Study With a Personalized NeoAntigen Cancer Vaccine Combined With Anti-PD-1 in Metastatic Melanoma
Brief Title: A Personalized NeoAntigen Cancer Vaccine Combined With Anti-PD-1 in Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, pfkchenxiang, Chen Xiang, Principal Investigator，Clinical Professor，Vice-President, Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYM001
Record Dates: First submitted 2019-07-26; First posted 2019-08-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Melanoma (Skin)
Keywords: Melanoma, Metastasis
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Peptides; spartalizumab; toripalimab; regramostim; Imiquimod

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/Treatment (Experimental): Personalized NeoAntigen Cancer Vaccine- Neo-Vac-Mn (peptides + rhGM-CSF+anti-PD1+Imiquimod 5% Topical Cream)
  NeoAntigen peptides:4 x 2 mg the total peptides given on days 84，87，91，98，105，133，and 161
  Anti-PD-1 Toripalimab: 3mg/kg, ivgtt, Q2w
  rhGM-CSF: 3μg/kg given on Days 81，82，83，95，96，97，102，103，104，130，131，132，158，159，and 160
  Imiquimod 5% Topical Cream:topical application on the injection site 6 hours before each NeoAntigen peptides injection
  Interventions: Drug: Peptide; Drug: Anti-PD-1; Drug: rhGM-CSF; Drug: Imiquimod 5% Topical Cream

INTERVENTIONS:
Drug: Peptide — 4 x 3 mg all the peptides given on days 84，87，91，98，105，133，and 161
  Other Names: NeoAntigen peptides
Drug: Anti-PD-1 — 3mg/kg, ivgtt, Q2w
  Other Names: Toripalimab
Drug: rhGM-CSF — 3μg/kg given on Days 81，82，83，95，96，97，102，103，104，130，131，132，158，159，and 160
Drug: Imiquimod 5% Topical Cream — topical application on the injection site 6 hours before each NeoAntigen peptides injection

SUMMARY:
This study assessed the safety and efficacy of individualized new antigen cancer vaccine combined with Programmed Cell Death Protein 1（PD1） inhibitor Toripalimab in the treatment of metastatic cutaneous melanoma. Melanoma is the most malignant skin neoplasm. Immunotherapy is the main treatment at present. PD1 is an immunological checkpoint and the inhibitors can reduce the immune escape of tumors, enhance T cell function and kill tumors. At present, PD1 antibody is the representative drug of immunotherapy, but the overall efficiency of its single drug treatment of acral melanoma is still low, and the combined treatment can significantly improve the efficiency. Melanoma has a high mutation load, which makes each patient have mutations specific to individual patients and tumors (changes in genetic material). These mutations lead to tumour cells producing proteins that are distinct from those of the body's own cells. These proteins used in vaccines may cause a strong immune response, which may help participants' bodies fight against any cancer cells that may lead to future recurrence of melanoma. Inhibition of PD1 can enhance the activity of T cells and form T cells with sustained killing activity. Tumor vaccines activate human Antigen Presenting Cells (APC) by injecting tumor antigens and adjuvants, and then activate T cells by APC to produce specific killing T cells. Therefore, the combination of "tumor vaccine + PD1 inhibitor" can produce effective specific killing and sustained activation of T cells, and prevent the establishment of inhibitory tumor microenvironment by tumor cells. The study will examine the safety and efficiency of the combined therapy at different time points and assess whether there is an immune response in the patient's peripheral blood and tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must meet the following criteria on screening examination to be eligible to participate in the study:
2. Patient is willing and able to give written informed consent.
3. Age ≥ 18 years, ≤75 years
4. Pathologically confirmed, clinically evident (by physical examination or radiographic imaging) stage IIIDN3c、IVM1a、M1b、M1c cutaneous melanoma.
5. Lesions that can be measured，and at least one lesion that can be used to evaluate the efficacy of immunotherapy;Multiple biopsies are available for lesions.
6. Patient is agreeable to allow tumor、normal tissue samples and blood samples to be submitted for genomic/complete exome/transcriptional sequencing；
7. ECOG score is 0 or 1
8. Life expectancy >6 months
9. Normal organ and bone marrow function as defined below:

   Leukocytes ≥ 3,500/mcL Absolute lymphocyte count > 800/mcL Absolute neutrophil count > 1,500/mcL Platelets > 100,000/mcL Hemoglobin > 10.0 g/dL Total serum bilirubin < 1.0 x institutional upper limit of normal AST (SGOT)/ALT (SGPT) < 2.0 x institutional upper limit of normal Serum creatinine< 1.5 x institutional upper limit of normal
10. Women of childbearing potential (WOCBP) must have a negative pregnancy test before entering the trial and within 7 days prior to start of study medication.
11. Female patients enrolled in the study, short-term have no fertility plan and must agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy.
12. Male patients must agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy.
13. Good compliance, able to follow research protocols and follow-up procedures.

Exclusion Criteria:

1. Patients who meet any of the following criteria will not be eligible for this study.
2. Uveal or mucosal melanoma；
3. Patients who received immunotherapy or other targeted cancer therapy within 4 weeks (including, but not limited to: IL-2, CTLA-4 blockade, PD-1/PD-L1 blockade, but exception of INF-α given as adjuvant treatment)
4. Previous bone marrow or stem cell transplant
5. History of severe allergic reactions attributed to any vaccine therapy
6. Active, known, or suspected autoimmune disease with the exception of vitiligo, type 1 diabetes, or psoriasis not requiring systemic treatment.
7. Use of a non-oncology vaccine therapy for prevention of infectious diseases (up-to) 4 weeks prior to enrollment to the study. Patients may not receive any non-oncology vaccine therapy during the period of NeoVax administration and until at least 8 weeks after the last dose of study therapy
8. In an immunosuppressive stage or immunosuppressive drugs were used systematically within 2 weeks.
9. Patients with long-term use of glucocorticoids or with experimental anti-tumor drugs
10. Active bacterial or fungal infections identified clinically (>= level 2 of NCI-CTC edition 3);
11. Known chronic infections with HIV, hepatitis B or C
12. Known active or latent tuberculosis infection
13. A history of idiopathic pulmonary fibrosis and organized pneumonia, or active pneumonia on chest computed tomography.
14. Complicated with other tumors, except for cervical cancer in situ and basal cell carcinoma five years ago.
15. Severe coronary or cerebrovascular disease, or other diseases that the investigators considered should to be exclusion;
16. Drug abuse, Clinical, psychological or social factor result in affecting informed consent or research implementation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-21 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing adverse events | up to a maximum of 252 days
  Number of participants experiencing clinical and laboratory adverse events (AE)
Number of Patients with Complete Remission Rate | up to a maximum of 252 days
  Number of Patients with Complete Remission Rate（CRR）
Number of Patients with Progressive Disease | up to a maximum of 252 days
  Number of Patients with Progressive Disease（PD）
Number of Patients with Partial Response | up to a maximum of 252 days
  Number of Patients with Partial Response（PR）

SECONDARY OUTCOMES:
Monitoring of cellular immune response | up to a maximum of 252 days
  the immune response of serum and tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Chen, Doctor's, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ott PA, Hu Z, Keskin DB, Shukla SA, Sun J, Bozym DJ, Zhang W, Luoma A, Giobbie-Hurder A, Peter L, Chen C, Olive O, Carter TA, Li S, Lieb DJ, Eisenhaure T, Gjini E, Stevens J, Lane WJ, Javeri I, Nellaiappan K, Salazar AM, Daley H, Seaman M, Buchbinder EI, Yoon CH, Harden M, Lennon N, Gabriel S, Rodig SJ, Barouch DH, Aster JC, Getz G, Wucherpfennig K, Neuberg D, Ritz J, Lander ES, Fritsch EF, Hacohen N, Wu CJ. An immunogenic personal neoantigen vaccine for patients with melanoma. Nature. 2017 Jul 13;547(7662):217-221. doi: 10.1038/nature22991. Epub 2017 Jul 5. PMID 28678778
- [Result] Sahin U, Derhovanessian E, Miller M, Kloke BP, Simon P, Lower M, Bukur V, Tadmor AD, Luxemburger U, Schrors B, Omokoko T, Vormehr M, Albrecht C, Paruzynski A, Kuhn AN, Buck J, Heesch S, Schreeb KH, Muller F, Ortseifer I, Vogler I, Godehardt E, Attig S, Rae R, Breitkreuz A, Tolliver C, Suchan M, Martic G, Hohberger A, Sorn P, Diekmann J, Ciesla J, Waksmann O, Bruck AK, Witt M, Zillgen M, Rothermel A, Kasemann B, Langer D, Bolte S, Diken M, Kreiter S, Nemecek R, Gebhardt C, Grabbe S, Holler C, Utikal J, Huber C, Loquai C, Tureci O. Personalized RNA mutanome vaccines mobilize poly-specific therapeutic immunity against cancer. Nature. 2017 Jul 13;547(7662):222-226. doi: 10.1038/nature23003. Epub 2017 Jul 5. PMID 28678784